CLINICAL TRIAL: NCT05483699
Title: Comparison of the Efficiency of Three Different Methods in Reducing Pain and Fear in Children During Intravenous Cannulation: A Randomised Controlled Study
Brief Title: Efficiency of Three Different Methods in Reducing Pain in Children During Intravenous Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, DİDEM COŞKUN ŞİMŞEK, Principal Investigator, Firat University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: intravenous cannulation
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Child, Only
Keywords: Blowing bubbles; child; fear; kaleidoscope; pain; squeezing soft ball
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Squeezing a ball during intravenous cannulation reduces the child's pain and fear. (Experimental): The soft ball has a diameter of about 8-10 cm and can return to its old form when it is squeezed.
  Interventions: Other: Squeezing a ball
- Using a kaleidoscope during intravenous cannulation reduces the child's pain and fear. (Experimental): Kaleidoscope includes shapes of flowers and mirrors in the shape of triangle placed with an angle of 600. While rotating one of the cylinders, various shapes and colourful eyes are formed when viewed with one eye. When the kaleidoscope is rotated, the patterns look different all the time because the colourful parts are moving, attracting the child's attention.
  Interventions: Other: Kaleidoscope
- Blowing bubbles during intravenous cannulation reduces the child's pain and fear. (Experimental): Children in this group were shown bubble blower before intravenous cannulation and they were shown how bubbles formed and how to blow. Children blew bubbles during intravenous cannulation
  Interventions: Other: Blowing bubbles

INTERVENTIONS:
Other: Squeezing a ball — The children in the squeezing soft ball group were given the ball before the procedure. They were told to squeeze and loosen the ball with the hand that was not used for the procedure while intravenous cannula was being inserted.
  Arms: Squeezing a ball during intravenous cannulation reduces the child's pain and fear.
Other: Blowing bubbles — The children in the blowing bubble group were shown the bubble blower before intravenous cannulation and they were told how bubbles were formed and how they would blow. During intravenous cannulation, the child blew the blower
  Arms: Blowing bubbles during intravenous cannulation reduces the child's pain and fear.
Other: Kaleidoscope — Children in the Kaleidoscope group were given the kaleidoscope before intravenous cannulation and they were shown how to use it. The children were told to look at the kaleidoscope during the procedure until the procedure ended
  Arms: Using a kaleidoscope during intravenous cannulation reduces the child's pain and fear.

SUMMARY:
Purpose: This study investigates the effects of squeezing a soft ball, using a kaleidoscope, or blowing bubbles during intravenous cannulation on the pain and fear of children between the ages of 4 and 6.

Design and Methods: This study is a randomised controlled study. In the study, there were 30 children in the soft ball group, 30 children in the kaleidoscope group, 30 children in the bubbles group, and 30 children in the control group.

DETAILED DESCRIPTION:
15 minutes before the intravenous cannulation procedure, the second researcher interviewed the parents and the children in squeezing soft ball, kaleidoscope, blowing bubbles and control groups separately and filled in descriptive information form and Children's Fear Scale. After randomization, the second researcher, the child and the parent went to the blood collection room for the procedure. Children in the Kaleidoscope group were given the kaleidoscope before intravenous cannulation and they were shown how to use it. The children were told to look at the kaleidoscope during the procedure until the procedure ended. The children in the squeezing soft ball group were given the ball before the procedure. They were told to squeeze and loosen the ball with the hand that was not used for the procedure while intravenous cannula was being inserted. The children in the blowing bubble group were shown the bubble blower before intravenous cannulation and they were told how bubbles were formed and how they would blow. During intravenous cannulation, the child blew the blower. Routine procedures were applied on the children in the control group without any interventions. Inserting the intravenous cannula took 3-5 minutes. The procedure was carried out in the same room by the same nurse for four of the groups. After the intravenous cannulation procedure ended, a researcher and parents filled in Faces Pain Scale-Revised and Children's Fear Scale separately and independently to find out the level of pain and fear experienced by the child during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* parents who agreed to participate in the study

Exclusion Criteria:

* visually impaired child
* mentally retarded child
* speech impaired children

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
assessing fear during intravenous cannula | 3-5 minutes.
  Children's Fear Scale: The scale was developed by McMurtry et al. to find out the anxiety levels of children between 4 and 10 years of age (McCarthy et al., 2010). There are five face pictures in the scale. Anxiety level is scored between "0 and 4". 0 indicates "no anxiety", while a scared face is scored 4 and indicates "too much anxiety".
  After the intravenous cannulation procedure ended, a researcher and parents filled Children's Fear Scale separately and independently to find out fear experienced by the child during the procedure.
assessing pain during intravenous cannula | 3-5 minutes.
  Faces Pain Scale-Revised: The scale developed by Bieri et al. is used to evaluate the pain levels of children between the ages of 4 and 17 (Bieri, Reeve, Champion, Addicoat, & Ziegler, 1990). There are pictures of 6 faces in the scale. Level of pain is evaluated as "0,2,4,6,8,10". The face on the leftmost side is given a score of 0 and interpreted as "no pain", while the face on the rightmost side is given a score of 10 and interpreted as "a lot of pain". Pain severity increases as score increases.
  After the intravenous cannulation procedure ended, a researcher and parents filled Faces Pain Scale separately and independently to find out pain experienced by the child during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Coşkun Şimşek, Elâzığ, Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No